CLINICAL TRIAL: NCT03605407
Title: Effects of the Visit Prior to Hospital Admission on Anxiety, Depression and Satisfaction of Patients in an Intensive Care Unit
Brief Title: Patients Visit Prior to Hospital Admission & Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, PhD, MSc, PT, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ICU-visit-patients
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Anxiety; Depression; Intensive Care Unit Syndrome
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patient receiving one visit prior to hospital admission
  Interventions: Other: Patient visit prior to hospital admission
- Control group (No Intervention): Patient without receiving one visit prior to hospital admission

INTERVENTIONS:
Other: Patient visit prior to hospital admission — Patient and family receiving one visit prior to hospital admission for surgery
  Arms: Experimental group

SUMMARY:
The present study evaluates the effects of the visit prior to hospital admission on anxiety, depression and satisfaction of patients in an intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient at hospital admission for surgery

Exclusion Criteria:

* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | Change from Baseline anxiety and depression at 90 days
  Anxiety subscale range from 0 to 21. Depression subscale range from 0 to 21. Higher values represent a worse outcome (higher depression or anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gonzalez-Martin S, Becerro-de-Bengoa-Vallejo R, Angulo-Carrere MT, Iglesias ME, Martinez-Jimenez EM, Casado-Hernandez I, Lopez-Lopez D, Calvo-Lobo C, Rodriguez-Sanz D. Effects of a visit prior to hospital admission on anxiety, depression and satisfaction of patients in an intensive care unit. Intensive Crit Care Nurs. 2019 Oct;54:46-53. doi: 10.1016/j.iccn.2019.07.001. Epub 2019 Jul 26. PMID 31358482